CLINICAL TRIAL: NCT07287449
Title: A Multi-Center, Prospective Historically Controlled Clinical Trial Comparing the Safety and Effectiveness of Triadyme-C to a Total Disc Replacement Control Cohort in the Treatment of Symptomatic Cervical Disc Disease (SCDD) at a Single Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dymicron (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-22012
Record Dates: First submitted 2025-12-12; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cervical Disc Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Safety and Effectiveness of Triadyme-C (Experimental): To evaluate the safety and effectiveness of the Triadyme-C device in comparison to other approved TDRs in the treatment of symptomatic cervical disc disease (SCDD) in subjects who are symptomatic at only a single level from C3 to C7 that are unresponsive to conservative management.
  Interventions: Device: Triadyme-C

INTERVENTIONS:
Device: Triadyme-C — Triadyme-C Cervical Total Disc Replacement

SUMMARY:
A multicenter, prospective, historically controlled study to evaluate the safety and effectiveness of the Triadyme-C device in comparison to other approved TDRs in the treatment of symptomatic cervical disc disease (SCDD) in subjects who are symptomatic at only a single level from C3 to C7 that are unresponsive to conservative management.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject, age ≥21.
2. Diagnosis of radiculopathy or myeloradiculopathy of the cervical spine, with pain, paresthesia or paralysis in a specific nerve root distribution C3 through C7, including at least one of the following:

   1. Neck and/or arm pain (at least 30 mm on the 100 mm visual analogue scale [VAS] scale).
   2. Decreased muscle strength of at least one level on the clinical evaluation 0 to 5 scale.
   3. Abnormal sensation including hyperesthesia or hypoesthesia; and/or
   4. Abnormal reflexes.
3. Symptomatic at a single level from C3 to C7.
4. Radiographically determined pathology at the level to be treated correlating to primary symptoms including at least one of the following:

   1. Decreased disc height on radiography, computed tomography (CT), or magnetic resonance imaging (MRI) in comparison to a normal adjacent disc.
   2. Degenerative spondylosis on CT or MRI.
   3. Disc herniation on CT or MRI.
5. Neck Disability Index (NDI) Score ≥ 30 (out of 100).
6. Unresponsive to non-operative, conservative treatment (e.g., rest, heat, electrotherapy, physical therapy, chiropractic care and/or analgesics) for:

   1. At least six weeks from radiculopathy or myeloradiculopathy symptom onset; or
   2. Have the presence of progressive symptoms or signs of nerve root/spinal cord compression despite continued non-operative conservative treatment.
7. Appropriate for treatment using an anterior surgical approach.
8. Reported to be medically cleared for surgery.
9. Reported to be physically and mentally able and willing to comply with the Protocol, including the ability to read and complete required forms and willing and able to adhere to the scheduled follow-up visits and requirements of the Protocol.
10. Written informed consent provided by subject.

Exclusion Criteria:

1. Have an active systemic infection or infection at the operative site.
2. Have a history of or anticipated treatment for active systemic infection, including HIV or Hepatitis C.
3. Have more than one immobile vertebral level between C1 to C7 from any cause including but not limited to congenital abnormalities and osteoarthritic "spontaneous" fusions.
4. Have previous trauma to the C3 to C7 levels resulting in significant bony or disco-ligamentous cervical spine injury.
5. Prior attempted or completed cervical spine surgery at any cervical level, except (1) a minimally invasive decompression that did not de-stabilize the segment upon flexion/extension or (2) a successful single-level anterior cervical fusion at non-index level (greater than 6 months prior to scheduled surgical treatment).
6. Have axial neck pain in the absence of other symptoms of radiculopathy or myeloradiculopathy justifying the need for surgical intervention.
7. Have disc height less than 3 mm as measured from the center of the disc in a neutral position.
8. Evidence of symptomatic moderate to severe facet joint degeneration or disease where the investigator feels this is a major contributor to the subject's pain as diagnosed by injection and imaging.
9. Have osteoporosis or is an increased risk of osteoporosis/osteopenia defined as a T-score less than -1.5 (i.e., -1.6, -1.7, etc.).

   1. The SCORE/MORES will be used to screen if a dual energy X-ray absorptiometry (DEXA) scan is required. If SCORE/MORES value ≥ 6, then a DEXA is required.
   2. An existing DEXA is allowed if completed within 12 months of subject surgery.
10. Have diabetes mellitus requiring daily insulin management.
11. Have severe myelopathy to the extent that the patient is wheelchair bound.
12. Have Paget's disease, osteomalacia or any other metabolic bone disease other than osteoporosis, which is addressed above (i.e., Exclusion #9).
13. Have active malignancy that includes a history of any invasive malignancy (except non-melanoma skin cancer) unless the subject had been treated with curative intent and there has been no clinical signs or symptoms of the malignancy for at least five years.
14. Have tumor as source of symptoms.
15. Have Symptomatic Cervical Degenerative Disc Disease (SDDD) or significant cervical spondylosis at two or more levels.
16. Have spondylolysis.
17. Have arachnoiditis.
18. Have marked cervical instability on resting (neutral) lateral or flexion-extension radiographs demonstrated by:

    1. Translation ≥ 3.5 mm, and/or
    2. Greater than 11° angular difference to that of either adjacent level.
19. Have a known allergy to implant materials (titanium, Ti-6Al-4V alloy, TiC, or SnCoCrMo alloy).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical Success | 24 months
  At least 15-point improvement in NDI Score (out of 100) compared with baseline.
Composite Clinical Success | 24 months
  Maintenance or improvement in neurological status (motor and sensory only) compared to baseline as adjudicated by the CEC.
Composite Clinical Success | 24 months
  No secondary surgical interventions (revision, removal, re-operation, supplemental fixation) at the index level.
Composite Clinical Success | 24 months
  Absence of serious device-related adverse events, as adjudicated by the CEC.

SECONDARY OUTCOMES:
Clinically Significant Improvement | 6 weeks
  Clinically significant improvement in one or more radicular symptoms or myelopathy at each timepoint compared to baseline.
Clinically Significant Improvement | 3 months
  Clinically significant improvement in one or more radicular symptoms or myelopathy at each timepoint compared to baseline.
Clinically Significant Improvement | 6 months
  Clinically significant improvement in one or more radicular symptoms or myelopathy at each timepoint compared to baseline.
Clinically Significant Improvement | 12 months
  Clinically significant improvement in one or more radicular symptoms or myelopathy at each timepoint compared to baseline.
Clinically Significant Improvement | 24 months
  Clinically significant improvement in one or more radicular symptoms or myelopathy at each timepoint compared to baseline.